CLINICAL TRIAL: NCT01390285
Title: Effect of Transcutaneous Electrical Nerve Stimulation in Relation to Central Sensitization in Patients With Osteoarthritis of the Knee: a Randomized Controlled Clinical Trial.
Brief Title: Transcutaneous Electrical Nerve Stimulation in Relation to Central Sensitization in Osteoarthritis of the Knee
Acronym: TENSSENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: David Beckwée, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tenssens
Record Dates: First submitted 2011-04-13; First posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TENS (Experimental)
  Interventions: Device: Transcutaneous electric nerve stimulation
- Sham TENS (Sham Comparator)
  Interventions: Device: sham transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electric nerve stimulation — The subjects that enter the TENS-group will be asked to apply the TENS therapy for at least 40 minutes continuously per day. The parameters of the current will not be changed during the study (pulse: 250 µsec; internal frequency: 100Hz; burst frequency 3 Hz; intensity: until an unpleasant but not painful sensation is acquired).
  Arms: TENS
Device: sham transcutaneous electrical nerve stimulation — The patients that are assigned to the sham TENS will receive an inactive placebo TENS therapy using a nonfunctional unit that appears to work but provides no stimulus.
  Arms: Sham TENS

SUMMARY:
Background

Central sensitization has recently been documented in patients with knee osteoarthritis. So far, the presence of central sensitization has not been considered as a confounding factor in studies assessing the pain inhibitory effect of TENS on osteoarthritis of the knee.

Purpose

First, to explore the pain inhibitory effect of burst TENS in OAk patients. Second, to explore the prognostic value of central sensitization on the pain inhibitory effect of TENS in Oak patients.

Methods

Patients with knee pain due to OAk will be recruited through advertisements in local media. Temporal summation, before and after a heterotopic noxious conditioning stimulation, will be measured. In addition, pain on a numeric rating score and WOMAC subscores for pain and function will be assessed. Patients will be randomly allocated to one of two treatment groups (TENS, sham TENS). Follow-up measurements will be scheduled after a period of 6 and 12 weeks.

Discussion/ conclusion

TENS influences pain through the electrical stimulation of low-threshold A-beta cutaneous fibers. The responsiveness of central pain-signaling neurons of OAk patients who are centrally sensitized may be augmented to the input of these electrical stimuli. This would encompass an adverse therapy effect of TENS. Therefore it might be interesting to identify a subgroup of symptomatic OAk patients, ie. non-sensitized patients, who are likely to benefit from burst TENS.

ELIGIBILITY:
Inclusion Criteria:

* To be included, patients need to be over 50 years old.
* All should have osteoarthritis in at least one knee fulfilling the American College of Rheumatology classification criteria and report peak knee pain over the last 24 h of more than 3 on a Numeric Rating Score (0-10 scale).

Exclusion Criteria:

* Patients are excluded if they have had a knee surgery or intra-articular corticosteroid injection within 6 months
* Current or past (within 4 weeks) oral corticosteroid use
* A history of knee joint replacement or tibial osteotomy
* Contraindications to burst TENS (pacemakers, epilepsy, dermatological conditions, abnormal sensation in the knees, pregnancy) or if they are unable to apply TENS independently

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Overall average knee pain | after 6 and 12 weeks
  numeric rating score

SECONDARY OUTCOMES:
Change from baseline in self reported knee pain and difficulty with physical function (WOMAC) | baseline - 6 weeks
Change from baseline in self reported knee pain and difficulty with physical function (WOMAC) | baseline - 12 weeks

REFERENCES:
- [Derived] Beckwee D, De Hertogh W, Lievens P, Bautmans I, Vaes P. Effect of tens on pain in relation to central sensitization in patients with osteoarthritis of the knee: study protocol of a randomized controlled trial. Trials. 2012 Feb 21;13:21. doi: 10.1186/1745-6215-13-21. PMID 22353582